CLINICAL TRIAL: NCT04321798
Title: A Novel, Theory Based Intervention to Promote Engagement in Physical Activity in Early Rheumatoid Arthritis (PEPA-RA): Proof of Concept Study
Brief Title: Promoting Engagement in Physical Activity in Early Rheumatoid Arthritis: Proof of Concept Study
Acronym: PEPA-RA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the West of England (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HAS.17.04.144
Record Dates: First submitted 2019-01-25; First posted 2020-03-25 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Rheumatoid Arthritis
Keywords: fatigue; physical activity; quality of life; function
MeSH Terms: conditions — Arthritis, Rheumatoid; Fatigue; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physical Activity (Experimental): Promoting Engagement in Physical Activity
  Interventions: Behavioral: Physical Activity

INTERVENTIONS:
Behavioral: Physical Activity — Four group sessions and one individual session delivered over a period of 12 weeks in a primary care setting. Each session includes patient education and support for behaviour change as well as a supervised practical exercise component. The intervention is based upon a combination of self-determination theory and COM-B framework (capability, opportunity, motivation and behaviour) and employs motivational interviewing techniques.

SUMMARY:
People with rheumatoid arthritis have indicated that they would like better support to remain physically active following diagnosis and would welcome a physical activity programmes delivered outside of a secondary care setting by a physiotherapist. With patient input, and based upon previous research in other long term conditions, a physical activity intervention was developed by the researchers for delivery by musculoskeletal physiotherapists in a primary care setting.

This proposed proof of concept study will investigate the new intervention and inform a future randomised controlled pilot trial. Four Band 6 musculoskeletal physiotherapists will be trained to deliver the intervention. Subsequently up to 32 patients with a recent diagnosis of rheumatoid arthritis (6 -24 months previously) will be recruited. Each physiotherapist will deliver the 12-week intervention package to a group of 6-8 participants. The participants will be asked to complete some outcome measures at the beginning of the 12-week intervention and again at the end.

Following the 12-week programme some of the patients will be asked what they thought of the programme and the outcome measures and whether they have any suggestions for improvement. Those that did and did not complete the programme will be included to ensure a wide range of views. The treating physiotherapists will also be asked about their experiences of delivering the programme as well as what they thought of the training.

Based upon these findings the programme will be refined and if appropriate further funding sought to carry out a pilot randomised controlled trial.

DETAILED DESCRIPTION:
A novel, theory based intervention to promote engagement in physical activity in early rheumatoid arthritis (PEPA-RA): proof of concept study.

People with rheumatoid arthritis (RA) do less physical activity (PA) than the general population and this is associated with work disability and reduced physical function. High intensity training and supervised exercise can improve physical function in RA, while PA decreases chronic inflammation and reduces pain, all without adversely affecting disease activity. Despite the benefits, patients do not maintain exercise beyond the supervised intervention and benefits are not maintained.

People with RA report a range of barriers to PA and are often reluctant to participate for fear of exacerbating their symptoms. It is therefore essential that they are provided with appropriate support to overcome these barriers soon after diagnosis, in order to optimise PA, minimise inappropriate health beliefs and prevent unnecessary reductions in function. Patients have also expressed a desire for more information relating to exercise.

Physiotherapists are best placed to provide this support as their approach is person-centred, taking into account the individual's health and wellbeing needs and supporting self-management through patient education and the facilitation of behaviour change. Whilst the National Institute for Health and Care Excellence (NICE) guidelines indicate that people with RA should have access to specialist physiotherapy to encourage regular PA this rarely occurs in practice with a third of patients waiting over a year for physiotherapy. The British Society of Rheumatology suggests that conversations regarding health promotion, including PA, need to occur early in the patient pathway and are best delivered via primary care.

To explore the opinions of people with RA in relation to support for PA programmes the investigators carried out focus groups. Based upon these findings, in combination with existing evidence and input from patient research partners, the researchers designed an intervention for delivery in a primary care setting for people with recently diagnosed RA. The focus group participants were in agreement that the intervention should be delivered in an accessible location within their local community. The intervention is informed by a theoretical framework for health behaviour change. The overall purpose of this new intervention is to support long term engagement with PA in order to optimise maintenance of physical function. The researchers plan to investigate the effectiveness of the intervention in a future trial, but initially need to carry out a proof of concept study.

Aim: to test the feasibility of a novel intervention and inform a future randomised controlled pilot trial of the refined intervention.

Objectives:

* To explore acceptability and feasibility of the intervention to patients and physiotherapists including the format, delivery method and location, content and support materials.
* To explore the acceptability of the physiotherapists training package.
* To refine the physiotherapists training and patient intervention packages.
* To determine acceptability and completeness of all the outcome measures. Up to 36 people with a recent diagnosis of RA will be recruited to take part in one of 4 PA intervention groups with 6-8 participants per group.

Patients will be recruited from secondary care Rheumatology outpatient clinics. Nursing staff will receive a familiarisation session about the study and be encouraged to briefly discuss it with all recently diagnosed RA patients. If patients express interest in taking part, a full information sheet will be provided. Those declining the trial will be offered a copy of the 'Keep Moving' booklet published by Arthritis Research UK. Where possible, reasons for declining will be gathered.

Those interested will receive a brief telephone screening interview at a time of their convenience (conducted by the Research Fellow). During the telephone call, patients will be given an opportunity to ask questions about the study. Patients who confirm verbally that they would like to enter the study will be referred to the physiotherapists delivering the intervention. Following screening and informed consent potential participants will be invited to enrol in the study. Written consent will be obtained when the patients attend for the initial session.

Four Band 6 musculoskeletal physiotherapists from primary care settings will be trained, via two half day workshops, to deliver the PA intervention.

Physiotherapist Training will be led by a musculoskeletal physiotherapist with experience of delivering similar interventions to groups of RA and OA patients, as well as practical experience of working in a regional rheumatology centre. They will be supported by a Rheumatology Clinical Specialist Physiotherapist as well as experts in the delivery of similar PA health behaviour change interventions. Following training the four physiotherapists will each deliver the intervention to a group of 6-8 people with a recent diagnosis of RA (diagnosed 6 months to 2 years prior to recruitment).

The intervention consists of four group sessions and one individual session delivered over a period of 12 weeks in a primary care setting. Each session includes patient education and support for behaviour change as well as a supervised practical exercise component. The intervention is based upon a combination of self-determination theory and COM-B framework (capability, opportunity, motivation and behaviour) and employs motivational interviewing techniques. Motivational interviewing has been used successfully by a range of health professionals to promote behaviour change. The combination of group and individualised sessions is intended to facilitate peer support (providing relatedness) and ensure that participants are provided with individual support to meet specific needs (enhancing autonomy and competence).

Week 0 and 2 (2 hours each): The group (n=6-8) intervention commences with 2 sessions to set and review goals, facilitate engagement and motivation, create an autonomy supportive environment and facilitate relatedness (connection with others 'like me').

Week 4 (45 mins): Individualised session at a location that is agreed between the patient and physiotherapist. This will be guided by the patient's goals as well as practicalities faced by the physiotherapist including insurance issues and travel time. Example locations for the individual session may include the patient's home, a community gym or swimming pool. Participants will be supported to identify community facilities for PA (opportunity). The individualised session will facilitate discussion of individual barriers to PA and identification of strategies to overcome them that may be unique to the individual and their setting. Patients will be given the opportunity to invite a supportive 'other' to attend this session.

Weeks 8 & 12 (90 mins/session): Group consolidation sessions include discussion on problem solving in relation to barriers and setbacks, as well as relapse prevention. Due to the flare-up and remission pattern of RA there are periods when continued PA at the usual level is not practicable; recovery strategies and re-engagement methods are thus incorporated into the intervention. These sessions will also include 30 minutes of supervised exercise.

Patients will be asked to complete a range of outcomes at baseline and 12 weeks. All participants will be asked to attend for one hour prior to the week 0 session commencing and remain for one hour after the week 12 session to allow time for completion of outcomes. The Research Fellow will oversee the completion of the outcome measures to reduce the risk of bias from the physiotherapist delivering the intervention. The purpose of including these outcomes within this 'proof of concept' study is to explore their acceptability to patients, as well as to provide an indication of the interventions potential for benefit. Acceptability of the outcomes package (primary and secondary outcomes) will be explored through the subsequent patient interviews (described below), as well as through the percentage of data that is analysable. Our patient research partner completed the baseline patient reported outcomes and reported that they only took 14 minutes. They felt that this would be acceptable to most participants in the study in addition to the completion of the objective measures. The secondary outcomes are those proposed for the future definitive study:

In addition to the intervention outcomes the following data will be collected:

* Reasons for declining to take participate in the intervention
* Patient attendance at each of the five sessions
* Adverse events - data collected by the treating physiotherapist based upon events occurring during the sessions as well as events reported by the patient to have occurred between sessions.
* Queries received by the research team from the treating physiotherapists will be logged.

Following the three-month intervention, qualitative semi-structured face to face individual interviews will be undertaken with the four physiotherapists to explore their views regarding the training and support provided; the method of delivery of the intervention including number of sessions and time between sessions; content of the intervention and any other issues relating to the training, the intervention or the future study that they deem important. The physiotherapists will be encouraged to keep a reflective diary throughout the intervention that they may refer to during the interview. The interviews will be carried out by a Research Associate who has not had previous involvement in the study.

Patients will be invited to participate in semi-structured interviews (approximately n=12 dependent upon data saturation), in order to explore their experiences of the intervention, the support material and outcome measures. They will also be asked about any other outcomes that they experienced as a result of the study and about any contact that they made with the rheumatology team during the study period. The aim will be to recruit 2-3 people from each intervention group to participate including representation from those that dropped out before week 12, males and females, and a range of ages. Where possible face to face interviews will be carried out, but if this is not convenient for the patients then telephone interviews will be offered. The Research Associate employed to carry out the interviews with the physiotherapists will also conduct the patient interviews.

Quantitative outcome data will be reported using descriptive statistics including the percentage of patients with analysable data.

Inductive thematic analysis will be carried out on the data from the physiotherapy and patient interviews. The findings will then be used to help refine the physiotherapist training and the intervention package. This information will ultimately inform the design of a future randomised controlled pilot trial.

ELIGIBILITY:
Inclusion Criteria:

Adults with RA diagnosed in the previous 6-24 months. Able to undertake a PA programme. Able to understand and speak English. Able to understand the purpose of the research Provides informed consent.

Exclusion Criteria:

Diagnosis of RA less than 6 months or more than 2 years previously. Unable to participate for medical reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-06-29 (Actual); Study Completion 2018-06-29 (Actual)

PRIMARY OUTCOMES:
Intervention Attendance | 12 weeks
  minimum 0 maximum 5; higher is better

SECONDARY OUTCOMES:
International Physical Activity Questionnaire - Short Form | 7 days
  scores are categorised as low, moderate or high; high is better
6-minute walk distance | 6 minutes
  Distance walked in 6 minutes, minimum is 0, no maximum. Higher is better
modified Health Assessment Questionnaire | 7 days
  measures function. Scores are categorised mild, moderate or severe. Mild is better.
Bristol Rheumatoid Arthritis Fatigue - Numerical Rating Scales | 7 days
  three scales covering severity, effect and coping all scored from 0-10 with 10 being worst
Self-efficacy for Exercise | 7-days
  0-100 with higher indicating better self efficacy
Motivation to exercise: Behavioural Regulation In Exercise Questionnaire version 2 | 7-days
  minimum 0 maximum 76; higher score is better
Generic quality of life: EuroQoL - EQ-5D-5L | day of completion
  Only the VAS values were reported with 0 minimum and 100 maximum; higher is better
Short Form 12 | 4 weeks
  physical and mental component subscales scored separately. Both range from 0 minimum to 100 maximum with higher scores indicating better outcome

CONTACTS AND LOCATIONS:
Locations (1):
- University of the West of England, Bristol, United Kingdom

IPD SHARING:
Plan to Share IPD: No
We do not have ethical approval to share IPD